CLINICAL TRIAL: NCT01499095
Title: 6-Month, Multicenter, Randomized, Open-label, Parallel-group Study Comparing the Efficacy and Safety of a New Formulation of Insulin Glargine and Lantus® Both in Combination With Oral Antihyperglycemic Drug(s) in Patients With Type 2 Diabetes Mellitus With a 6-month Safety Extension Period
Brief Title: Comparison of a New Formulation of Insulin Glargine With Lantus in Patients With Type 2 Diabetes on Basal Insulin With Oral Antidiabetic Therapy
Acronym: EDITION II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC11629; 2010-023770-39 (EudraCT Number); U1111-1118-6943 (Other: UTN)
Record Dates: First submitted 2011-12-16; First posted 2011-12-26 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOE901-U300 (Experimental)
  Interventions: Drug: HOE901-U300 (new formulation of insulin glargine)
- Lantus (Active Comparator)
  Interventions: Drug: Lantus (Insulin glargine)

INTERVENTIONS:
Drug: Lantus (Insulin glargine) — Lantus (HOE901-U100, insulin glargine 100 U/mL) SC injection once daily (evening) for 12 months in combination with oral antidiabetic drug(s). Dose titration seeking fasting plasma glucose 4.4-5.6 mmol/L (80 - 100 mg/dL).
  Other Names: Lantus
  Arms: Lantus
Drug: HOE901-U300 (new formulation of insulin glargine) — HOE901-U300 (new insulin glargine 300 units per milliliter [U/mL]) subcutaneous (SC) injection once daily (evening) for 12 months in combination with oral antidiabetic drug(s). Dose titration seeking fasting plasma glucose 4.4 - 5.6 millimole per liter (mmol/L) (80 - 100 milligram per deciliter [mg/dL]). After 6 months participants were proposed to participate to the administration substudy and to receive either HOE901-U300 once daily at intervals of 24 +/- 3 hours (adaptable dosing intervals) or to continue once daily injections of HOE901-U300 every 24 hours (fixed dosing intervals) up to Month 9.
  Arms: HOE901-U300

SUMMARY:
Primary Objective:

* To compare the efficacy of insulin glargine new formulation and Lantus in terms of change in Glycated Hemoglobin A1c (HbA1c) from baseline to endpoint (scheduled Month 6) in adult participants with type 2 diabetes mellitus

Secondary Objective:

* To compare the efficacy of insulin glargine new formulation and Lantus in terms of occurrence of nocturnal hypoglycemia

DETAILED DESCRIPTION:
The maximum study duration was up to approximately 58 weeks per participants, consisting of:

* up to 2 week screening period
* 6-month comparative efficacy and safety treatment period
* 6-month comparative safety extension period
* 4-week safety follow-up period in a subset of participants
* a 3-month administration substudy period starting after completion of the 6-month study period for participants willing to in a subset of participants randomized to HOE901-U300

ELIGIBILITY:
Inclusion criteria :

* Participants with type 2 diabetes mellitus
* Substudy inclusion criteria:

  * Completion of the 6-month study period in main study (Visit 10)
  * Randomized and treated with insulin glargine new formulation during the 6- month treatment period (Baseline - Month 6)

Exclusion criteria:

* Age less than (<) 18 years
* HbA1c <7.0% or greater than (>) 10% at screening
* Diabetes other than type 2 diabetes mellitus
* Less than 6 months on basal insulin treatment together with oral antihyperglycemic drug(s) and self-monitoring of blood glucose
* Participants using sulfonylurea in the last 2 months before screening visit
* Any contraindication to use of insulin glargine as defined in the national product label
* Use of insulin pump in the last 6 months before screening
* Initiation of new glucose-lowering medications in the last 3 months before screening visit
* History or presence of significant diabetic retinopathy or macular edema likely to require laser or injectable drugs or surgical treatment during the study period
* Pregnant or breast-feeding women or women who intend to become pregnant during the study period
* Substudy exclusion criteria:

  * Participant not willing to use the adaptable injection intervals on at least two days per week

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 811 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (213):
- United States (110):
  - Investigational Site Number 840517, Birmingham, Alabama
  - Investigational Site Number 840149, Chandler, Arizona
  - Investigational Site Number 840093, Glendale, Arizona
  - Investigational Site Number 840069, Phoenix, Arizona
  - Investigational Site Number 840110, Sun City, Arizona
  - Investigational Site Number 840068, Tempe, Arizona
  - Investigational Site Number 840015, Hot Springs, Arkansas
  - Investigational Site Number 840014, Little Rock, Arkansas
  - Investigational Site Number 840114, Little Rock, Arkansas
  - Investigational Site Number 840018, Mountain Home, Arkansas
  - Investigational Site Number 840027, Searcy, Arkansas
  - Investigational Site Number 840074, Anaheim, California
  - Investigational Site Number 840509, Bell Gardens, California
  - Investigational Site Number 840060, Greenbrae, California
  - Investigational Site Number 840057, La Jolla, California
  - Investigational Site Number 840003, La Mesa, California
  - Investigational Site Number 840026, Los Angeles, California
  - Investigational Site Number 840090, Mission Hills, California
  - Investigational Site Number 840099, Palm Springs, California
  - Investigational Site Number 840004, San Diego, California
  - Investigational Site Number 840124, Santa Barbara, California
  - Investigational Site Number 840012, Tustin, California
  - Investigational Site Number 840104, Colorado Springs, Colorado
  - Investigational Site Number 840128, Colorado Springs, Colorado
  - Investigational Site Number 840098, Denver, Colorado
  - Investigational Site Number 840518, Brandon, Florida
  - Investigational Site Number 840049, Daytona Beach, Florida
  - Investigational Site Number 840008, Jacksonville, Florida
  - Investigational Site Number 840520, Miami, Florida
  - Investigational Site Number 840025, New Port Richey, Florida
  - Investigational Site Number 840011, Ocoee, Florida
  - Investigational Site Number 840141, Palm Harbor, Florida
  - Investigational Site Number 840513, Pembroke Pines, Florida
  - Investigational Site Number 840528, Columbus, Georgia
  - Investigational Site Number 840050, Idaho Falls, Idaho
  - Investigational Site Number 840107, Nampa, Idaho
  - Investigational Site Number 840199, Chicago, Illinois
  - Investigational Site Number 840021, McHenry, Illinois
  - Investigational Site Number 840020, Springfield, Illinois
  - Investigational Site Number 840045, Avon, Indiana
  - Investigational Site Number 840077, Avon, Indiana
  - Investigational Site Number 840088, Avon, Indiana
  - Investigational Site Number 840089, Avon, Indiana
  - Investigational Site Number 840091, Avon, Indiana
  - Investigational Site Number 840130, Evansville, Indiana
  - Investigational Site Number 840142, Lafayette, Indiana
  - Investigational Site Number 840041, Paducah, Kentucky
  - Investigational Site Number 840034, Baltimore, Maryland
  - Investigational Site Number 840150, Baltimore, Maryland
  - Investigational Site Number 840031, Rockville, Maryland
  - Investigational Site Number 840063, Ann Arbor, Michigan
  - Investigational Site Number 840064, Dearborn, Michigan
  - Investigational Site Number 840094, Flint, Michigan
  - Investigational Site Number 840023, Southfield, Michigan
  - Investigational Site Number 840066, Eagan, Minnesota
  - Investigational Site Number 840081, Minneapolis, Minnesota
  - Investigational Site Number 840158, Biloxi, Mississippi
  - Investigational Site Number 840526, Chesterfield, Missouri
  - Investigational Site Number 840502, Butte, Montana
  - Investigational Site Number 840084, Fremont, Nebraska
  - Investigational Site Number 840085, Omaha, Nebraska
  - Investigational Site Number 840162, Las Vegas, Nevada
  - Investigational Site Number 840527, Las Vegas, Nevada
  - Investigational Site Number 840056, Las Vegas, Nevada
  - Investigational Site Number 840135, Summit, New Jersey
  - Investigational Site Number 840145, Toms River, New Jersey
  - Investigational Site Number 840087, Toms River, New Jersey
  - Investigational Site Number 840140, Calabash, North Carolina
  - Investigational Site Number 840139, Hickory, North Carolina
  - Investigational Site Number 840153, Hickory, North Carolina
  - Investigational Site Number 840047, Wilmington, North Carolina
  - Investigational Site Number 840024, Winston-Salem, North Carolina
  - Investigational Site Number 840065, Fargo, North Dakota
  - Investigational Site Number 840007, Cincinnati, Ohio
  - Investigational Site Number 840097, Columbus, Ohio
  - Investigational Site Number 840113, Dayton, Ohio
  - Investigational Site Number 840108, Maumee, Ohio
  - Investigational Site Number 840504, Eugene, Oregon
  - Investigational Site Number 840080, Medford, Oregon
  - Investigational Site Number 840148, Tipton, Pennsylvania
  - Investigational Site Number 840005, Uniontown, Pennsylvania
  - Investigational Site Number 840076, Greer, South Carolina
  - Investigational Site Number 840503, Simpsonville, South Carolina
  - Investigational Site Number 840048, Rapid City, South Dakota
  - Investigational Site Number 840028, Bristol, Tennessee
  - Investigational Site Number 840038, Chattanooga, Tennessee
  - Investigational Site Number 840042, Knoxville, Tennessee
  - Investigational Site Number 840160, Memphis, Tennessee
  - Investigational Site Number 840033, Memphis, Tennessee
  - Investigational Site Number 840022, Austin, Texas
  - Investigational Site Number 840078, Austin, Texas
  - Investigational Site Number 840519, Corpus Christi, Texas
  - Investigational Site Number 840001, Dallas, Texas
  - Investigational Site Number 840159, Dallas, Texas
  - Investigational Site Number 840115, Dallas, Texas
  - Investigational Site Number 840079, Houston, Texas
  - Investigational Site Number 840514, Houston, Texas
  - Investigational Site Number 840525, San Antonio, Texas
  - Investigational Site Number 840161, San Antonio, Texas
  - Investigational Site Number 840009, Draper, Utah
  - Investigational Site Number 840037, Orem, Utah
  - Investigational Site Number 840510, Salt Lake City, Utah
  - Investigational Site Number 840032, Chesapeake, Virginia
  - Investigational Site Number 840040, Norfolk, Virginia
  - Investigational Site Number 840095, Richmond, Virginia
  - Investigational Site Number 840072, Williamsburg, Virginia
  - Investigational Site Number 840134, Winchester, Virginia
  - Investigational Site Number 840523, Olympia, Washington
  - Investigational Site Number 840122, Walla Walla, Washington
  - Investigational Site Number 840019, Milwaukee, Wisconsin
- Canada (14):
  - Investigational Site Number 124024, Beamsville
  - Investigational Site Number 124025, Burlington
  - Investigational Site Number 124020, Calgary
  - Investigational Site Number 124019, Chilliwack
  - Investigational Site Number 124018, Coquitlam
  - Investigational Site Number 124016, Edmonton
  - Investigational Site Number 124014, Hamilton
  - Investigational Site Number 124004, Mirabel
  - Investigational Site Number 124026, Mississauga
  - Investigational Site Number 124002, Red Deer
  - Investigational Site Number 124013, Sherbrooke
  - Investigational Site Number 124011, Toronto
  - Investigational Site Number 124010, Victoria
  - Investigational Site Number 124022, Winnipeg
- Chile (12):
  - Investigational Site Number 152014, Osorno
  - Investigational Site Number 152012, Rancagua
  - Investigational Site Number 152005, Santiago
  - Investigational Site Number 152004, Santiago
  - Investigational Site Number 152003, Santiago
  - Investigational Site Number 152001, Santiago
  - Investigational Site Number 152013, Santiago
  - Investigational Site Number 152002, Santiago
  - Investigational Site Number 152007, Santiago
  - Investigational Site Number 152010, Santiago
  - Investigational Site Number 152006, Temuco
  - Investigational Site Number 152009, Valdivia
- Investigational Site Number 246001, Helsinki, Finland
- France (6):
  - Investigational Site Number 250001, La Rochelle
  - Investigational Site Number 250004, Le Creusot
  - Investigational Site Number 250005, Mantes-la-Jolie
  - Investigational Site Number 250002, Nantes
  - Investigational Site Number 250009, Strasbourg
  - Investigational Site Number 250003, Vénissieux
- Germany (6):
  - Investigational Site Number 276004, Künzing
  - Investigational Site Number 276003, Neumünster
  - Investigational Site Number 276008, Oberhausen
  - Investigational Site Number 276009, Pirna
  - Investigational Site Number 276007, Rehlingen-Siersburg
  - Investigational Site Number 276005, Wangen
- Hungary (10):
  - Investigational Site Number 348006, Baja
  - Investigational Site Number 348005, Budapest
  - Investigational Site Number 348003, Budapest
  - Investigational Site Number 348010, Budapest
  - Investigational Site Number 348009, Budapest
  - Investigational Site Number 348002, Eger
  - Investigational Site Number 348001, Makó
  - Investigational Site Number 348008, Mosonmagyaróvár
  - Investigational Site Number 348004, Pápa
  - Investigational Site Number 348007, Sátorlaljaújhely
- Mexico (8):
  - Investigational Site Number 484009, Acapulco
  - Investigational Site Number 484007, Guadalajara
  - Investigational Site Number 484008, Guadalajara
  - Investigational Site Number 484010, Guadalajara
  - Investigational Site Number 484006, Mexico City
  - Investigational Site Number 484001, Monterrey
  - Investigational Site Number 484003, Monterrey
  - Investigational Site Number 484004, Pachuca
- Portugal (2):
  - Investigational Site Number 620007, Matosinhos Municipality
  - Investigational Site Number 620004, Porto
- Romania (15):
  - Investigational Site Number 642008, Bacau
  - Investigational Site Number 642009, Brasov
  - Investigational Site Number 642003, Bucharest
  - Investigational Site Number 642001, Bucharest
  - Investigational Site Number 642002, Bucharest
  - Investigational Site Number 642014, Cluj-Napoca
  - Investigational Site Number 642006, Deva
  - Investigational Site Number 642011, Hunedoara
  - Investigational Site Number 642015, Iași
  - Investigational Site Number 642013, Oradea
  - Investigational Site Number 642010, Ploieşti
  - Investigational Site Number 642004, Reşiţa
  - Investigational Site Number 642007, Târgu Mureş
  - Investigational Site Number 642012, Timișoara
  - Investigational Site Number 642005, Timișoara
- Russia (13):
  - Investigational Site Number 643010, Moscow
  - Investigational Site Number 643007, Moscow
  - Investigational Site Number 643009, Saint Petersburg
  - Investigational Site Number 643006, Saint Petersburg
  - Investigational Site Number 643014, Saint Petersburg
  - Investigational Site Number 643008, Saint Petersburg
  - Investigational Site Number 643013, Saint Petersburg
  - Investigational Site Number 643004, Saint Petersburg
  - Investigational Site Number 643001, Saint Petersburg
  - Investigational Site Number 643011, Samara
  - Investigational Site Number 643002, Saratov
  - Investigational Site Number 643016, Ufa
  - Investigational Site Number 643005, Voronezh
- South Africa (10):
  - Investigational Site Number 710007, Benoni
  - Investigational Site Number 710006, Bloemfontein
  - Investigational Site Number 710014, Bloemfontein
  - Investigational Site Number 710002, Boksburg
  - Investigational Site Number 710003, Cape Town
  - Investigational Site Number 710010, Cape Town
  - Investigational Site Number 710008, eMkhomazi
  - Investigational Site Number 710001, Johannesburg
  - Investigational Site Number 710005, Pretoria
  - Investigational Site Number 710012, Somerset West
- Spain (6):
  - Investigational Site Number 724005, Barcelona
  - Investigational Site Number 724003, Málaga
  - Investigational Site Number 724006, Palma de Mallorca
  - Investigational Site Number 724001, Sabadell
  - Investigational Site Number 724002, Seville
  - Investigational Site Number 724004, Valancia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Yki-Jarvinen H, Bergenstal R, Ziemen M, Wardecki M, Muehlen-Bartmer I, Boelle E, Riddle MC; EDITION 2 Study Investigators. New insulin glargine 300 units/mL versus glargine 100 units/mL in people with type 2 diabetes using oral agents and basal insulin: glucose control and hypoglycemia in a 6-month randomized controlled trial (EDITION 2). Diabetes Care. 2014 Dec;37(12):3235-43. doi: 10.2337/dc14-0990. Epub 2014 Sep 5. PMID 25193531
- [Derived] Yale JF, Aroda VR, Charbonnel B, Sinclair AJ, Trescoli C, Cahn A, Bigot G, Merino-Trigo A, Brulle-Wohlhueter C, Bolli GB, Ritzel R. Glycaemic control and hypoglycaemia risk with insulin glargine 300 U/mL versus glargine 100 U/mL: A patient-level meta-analysis examining older and younger adults with type 2 diabetes. Diabetes Metab. 2020 Apr;46(2):110-118. doi: 10.1016/j.diabet.2018.10.002. Epub 2018 Oct 23. PMID 30366067
- [Derived] Bolli GB, Wysham C, Fisher M, Chevalier S, Cali AMG, Leroy B, Riddle MC. A post-hoc pooled analysis to evaluate the risk of hypoglycaemia with insulin glargine 300 U/mL (Gla-300) versus 100 U/mL (Gla-100) over wider nocturnal windows in individuals with type 2 diabetes on a basal-only insulin regimen. Diabetes Obes Metab. 2019 Feb;21(2):402-407. doi: 10.1111/dom.13515. Epub 2018 Oct 2. PMID 30160030
- [Derived] Bonadonna RC, Renard E, Cheng A, Fritsche A, Cali A, Melas-Melt L, Umpierrez GE. Switching to insulin glargine 300 U/mL: Is duration of prior basal insulin therapy important? Diabetes Res Clin Pract. 2018 Aug;142:19-25. doi: 10.1016/j.diabres.2018.03.041. Epub 2018 Apr 9. PMID 29649539
- [Derived] Yale JF, Pettus JH, Brito-Sanfiel M, Lavalle-Gonzalez F, Merino-Trigo A, Stella P, Chevalier S, Buzzetti R. The effect of concomitant DPPIVi use on glycaemic control and hypoglycaemia with insulin glargine 300 U/mL (Gla-300) versus insulin glargine 100 U/mL (Gla-100) in people with type 2 diabetes: A patient-level meta-analysis of EDITION 2 and 3. PLoS One. 2018 Jan 25;13(1):e0190579. doi: 10.1371/journal.pone.0190579. eCollection 2018. PMID 29370218
- [Derived] Yki-Jarvinen H, Bergenstal RM, Bolli GB, Ziemen M, Wardecki M, Muehlen-Bartmer I, Maroccia M, Riddle MC. Glycaemic control and hypoglycaemia with new insulin glargine 300 U/ml versus insulin glargine 100 U/ml in people with type 2 diabetes using basal insulin and oral antihyperglycaemic drugs: the EDITION 2 randomized 12-month trial including 6-month extension. Diabetes Obes Metab. 2015 Dec;17(12):1142-9. doi: 10.1111/dom.12532. Epub 2015 Sep 14. PMID 26172084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1250 participants were screened, of whom 439 participants were screen failure and 811 participants were randomized.
Pre-assignment Details: Following the main 6 month treatment period, eligible participants previously using HOE901-U300 were randomized (1:1) in a substudy and continued with fixed-dosing (every 24 hours) or started a adaptable-dosing (at intervals of 24 +/- 3 hours) regimen for 3 Months (Month 6 to 9).
Groups:
- HOE901-U300: HOE901-U300 (new insulin glargine 300 units per milliliter [U/mL]) subcutaneous (SC) injection once daily (evening) for 12 months in combination with oral antidiabetic drug(s).
- Lantus: Lantus (HOE901-U100, insulin glargine 100 U/mL) SC injection once daily (evening) for 12 months in combination with oral antidiabetic drug(s).
Period: Overall Study
Arm/Group | HOE901-U300 | Lantus
Started | 404 | 407
Treated | 403 | 406
Participated in Substudy | 89 (45 participants received adaptable dosing regimen and 44 participants received fixed dosing regimen) | 0
Modified Intent-to-Treat Population | 403 (Participants who received at least 1 dose of drug, had both baseline, at least 1 post-baseline data) | 405 (Participants who received at least 1 dose of drug, had both baseline, at least 1 post-baseline data)
Completed | 315 | 314
Not Completed | 89 | 93
Not completed — Randomized But Not Treated | 1 | 1
Not completed — Adverse Event | 12 | 7
Not completed — Lack of Efficacy | 2 | 1
Not completed — Protocol Violation | 6 | 7
Not completed — Received Rescue Therapy | 32 | 40
Not completed — Diverse Reasons | 22 | 25
Not completed — Lost to Follow-up | 6 | 4
Not completed — Insulin Dropped Below Authorized Dose | 0 | 5
Not completed — Hypoglycemia | 3 | 1
Not completed — Diagnosed With Type 1 Diabetes Mellitus | 2 | 1
Not completed — Change in Injection Schedule | 2 | 0
Not completed — Perceived Lack of Efficacy | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized population: all screened participants (who originally met inclusion criteria and signed informed consent) allocated to a treatment group and recorded in Interactive Voice/Web Response System (IVRS/IWRS) database, regardless of whether treatment was used or not. Participants were analyzed in treatment group to which they were randomized.
Groups:
- HOE901-U300: HOE901-U300 SC injection once daily for 12 months in combination with oral antidiabetic drug(s).
- Lantus: Lantus SC injection once daily for 12 months in combination with oral antidiabetic drug(s).
- Total: Total of all reporting groups
Arm/Group | HOE901-U300 | Lantus | Total
Number analyzed (Participants) | 404 | 407 | 811
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (9.1) | 58.5 (9.2) | 58.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 222 | 439
  Male | 187 | 185 | 372
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter] | 34.8 (6.6) | 34.8 (6.1) | 34.8 (6.4)
Duration of Diabetes [Median (Full Range); unit: years] — Number of participants analyzed for this baseline characteristics = 403 and 407 in HOE901-U300 and Lantus arm, respectively.
  years | 11.6 [1 to 54] | 11.7 [1 to 51] | 11.7 [1 to 54]
Basal Insulin Daily Dose [Mean (Standard Deviation); unit: units per kilogram] — Number of participants analyzed for this baseline characteristics = 378 and 382 in HOE901-U300 and Lantus arm, respectively.
  units per kilogram | 0.660 (0.221) | 0.681 (0.253) | 0.671 (0.238)
Glycated Hemoglobin A1c (HbA1c) [Number; unit: participants]
  Less Than (<) 8% | 144 | 146 | 290
  Greater Than or Equal to (>=) 8% | 260 | 261 | 521

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Month 6 Endpoint
Description: Only measurements performed before initiation of rescue therapy were considered in the analysis.
Time Frame: Baseline, Month 6
Population: Modified Intent-to-Treat population: all randomized participants who received at least (>=)1 dose, had baseline and >=1 post-baseline assessment of any efficacy variable, irrespective of compliance. Number of participants analyzed = participants with baseline and Week 6 HbA1c assessment. Missing data imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 386 | 392
percentage of hemoglobin | -0.57 (0.094) | -0.56 (0.093)
Statistical Analysis 1: Comparison: HOE901-U300 vs Lantus; Analysis was performed using an analysis of covariance (ANCOVA) model with treatment, strata of screening HbA1c (<8.0 and >=8.0%), and country as fixed effects and using the HbA1c baseline value as a covariate; Test type: Non-Inferiority or Equivalence — Stepwise closed testing approach was to assess non-inferiority and superiority sequentially: 1. Non-inferiority of HOE901-U300 vs Lantus: Upper bound of two-sided 95% confidence interval (CI) of difference between HOE901-U300 and Lantus on mITT population is <0.4%. 2. Superiority (only if non-inferiority has been demonstrated): Upper bound of two-sided 95% CI for difference in mean change in HbA1c from baseline to endpoint between HOE901-U300 and Lantus on mITT population is <0; Least Squares (LS) Mean difference = -0.01, 95% CI 2-sided [-0.139 to 0.119], Standard Error of Mean 0.066

2. Secondary Outcome: Percentage of Participants With At Least One Severe and/or Confirmed Nocturnal Hypoglycemia From Start of Week 9 to Month 6 Endpoint
Description: Nocturnal hypoglycemia was hypoglycemia that occurred between 00:00 and 05:59 hours (clock time), regardless the participant was awake or woke up because of the event. Severe hypoglycemia was an event that required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Confirmed hypoglycemia was an event associated with plasma glucose less than or equal to (<=) 3.9 mmol/L (70 milligram per deciliter [mg/dL]). Only measurements performed before initiation of rescue therapy were considered in the analysis.
Time Frame: Week 9 Up to Month 6
Population: Modified intent-to-treat population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 403 | 405
percentage of participants | 21.6 | 27.9
Statistical Analysis 1: Comparison: HOE901-U300 vs Lantus; A one-sided test (at alpha=0.025) for superiority of HOE901-U300 over Lantus was to be performed in case the non-inferiority of HOE901-U300 vs Lantus for the primary endpoint was demonstrated. Analysis was performed using Cochran-Mantel-Haenszel (CMH) method with treatment as a factor and stratified on strata of screening HbA1c (<8.0 and >=8.0%); Test type: Superiority or Other; p = 0.0380, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.61 to 0.99]

3. Secondary Outcome: Change in Average Preinjection Self-Monitored Plasma Glucose (SMPG) From Baseline to Month 6 Endpoint
Description: Preinjection SMPG was measured within 30 minutes prior to the injection of the study drug. Average was assessed by the mean of at least 3 SMPG calculated over the 7 days preceding the assessment visit. Only measurements performed before initiation of rescue therapy were considered in the analysis.
Time Frame: Baseline, Month 6
Population: mITT population. Missing data imputed using last observation carried forward. Number of participants analyzed = participants with baseline and Month 6 preinjection SMPG assessment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Groups:
- Lantus: Lantus SC injection once daily for 12 months on in combination with antidiabetic drug(s).
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 353 | 350
mmol/L | -0.56 (0.278) | -0.51 (0.275)
Statistical Analysis 1: Comparison: HOE901-U300 vs Lantus; Change in pre-injection SMPG was analysed using an ANCOVA model with treatment, strata of screening HbA1c (<8.0 and >=8.0%), and country as fixed effects and using the pre-injection SMPG baseline value as a covariate. A test for superiority of HOE901-U300 over Lantus was to be performed one-sided at level alpha = 0.025 if previous analysis for nocturnal hypoglycaemia was significant; Test type: Superiority or Other; p = 0.8279, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.438 to 0.350], Standard Error of Mean 0.201

4. Secondary Outcome: Change in Variability of Preinjection SMPG From Baseline to Month 6 Endpoint
Description: Preinjection SMPG was measured within 30 minutes prior to the injection of the study drug. Variability was assessed by the mean of co-efficient of variation calculated as 100 multiplied by (standard deviation/mean) over at least 3 SMPG measured during the 7 days preceding the assessment visit. Only measurements performed before initiation of rescue therapy were considered in the analysis.
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of mean
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 353 | 350
percentage of mean | -2.34 (1.425) | -0.53 (1.408)

5. Secondary Outcome: Percentage of Participants With HbA1c <7% at Month 6 Endpoint
Description: Only measurements performed before initiation of rescue therapy were considered in the analysis.
Time Frame: Month 6
Population: mITT Population. Number of participants analyzed = participants with Month 6 HbA1c assessment. Missing data imputed using last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 386 | 392
percentage of participants | 30.6 | 30.4

6. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Month 6 Endpoint
Description: Only measurements performed before initiation of rescue therapy were considered in the analysis.
Time Frame: Baseline, Month 6
Population: mITT Population. Number of participants analyzed = participants with baseline and Month 6 FPG assessment. Missing data imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 375 | 379
mmol/L | -1.03 (0.242) | -1.21 (0.241)

7. Secondary Outcome: Percentage of Participants With FPG <5.6 mmol/L (<100 mg/dL) at Month 6 Endpoint
Description: Only measurements performed before initiation of rescue therapy were considered in the analysis.
Time Frame: Month 6
Population: mITT Population. Number of participants analyzed = participants with Month 6 FPG assessment. Missing data imputed using last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 384 | 390
percentage of participants | 29.4 | 33.6

8. Secondary Outcome: Change in 8-Point SMPG Profiles Per Time Point From Baseline to Month 6 Endpoint
Description: Change in each time-point of 8-point SMPG profile: 03:00 hours (clock time) at night; before and 2 hours after breakfast; before and 2 hours after lunch; before and 2 hours after dinner; and at bedtime. Only measurements performed before initiation of rescue therapy were considered in the analysis.
Time Frame: Baseline, Month 6
Population: mITT population. Only participants from the mITT population with a value at baseline and at the specified timepoint were analyzed (represented by n=X, X in the category titles). Missing data imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 403 | 405
mmol/L
  03:00 at Night (n= 338, 328) | -0.56 (0.323) | -0.90 (0.321)
  Pre-breakfast (n= 347, 338) | -1.31 (0.221) | -1.81 (0.219)
  2 hours after breakfast (n= 341, 328) | -1.41 (0.331) | -1.82 (0.329)
  Pre-lunch (n= 344, 332) | -0.64 (0.300) | -1.12 (0.298)
  2 hours after lunch (n= 339, 328) | -1.02 (0.342) | -1.04 (0.340)
  Pre-dinner (n=347, 336) | -0.94 (0.327) | -0.69 (0.324)
  2 hours after dinner (n= 338, 327) | -0.69 (0.359) | -1.00 (0.357)
  Bedtime (n= 325, 303) | -0.99 (0.345) | -1.00 (0.343)

9. Secondary Outcome: Change in Daily Basal Insulin Dose From Baseline to Month 6 Endpoint
Description: Only measurements performed before initiation of rescue therapy were considered in the analysis.
Time Frame: Baseline, Month 6
Population: mITT Population. Number of participants analyzed = participants with Baseline and Month 6 basal insulin dose assessment. Missing data imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: U/kg
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 402 | 403
U/kg | 0.28 (0.021) | 0.17 (0.021)

10. Secondary Outcome: Change in Treatment Satisfaction Score Using The Diabetes Treatment Satisfaction Questionnaire (DTSQs) From Baseline to Month 6 Endpoint
Description: DTSQ is a validated measure to assess how satisfied participants with diabetes are with their treatment and how they perceive hyper- and hypoglycemia. It consists of 8 questions which are answered on a Likert scale from 0 to 6. DTSQ treatment satisfaction score is the sum of question 1 and 4-8 scores and ranges between 0 and 36, where higher scores indicate more treatment satisfaction. Only measurements performed before initiation of rescue therapy were considered in the analysis.
Time Frame: Baseline, Month 6
Population: mITT Population. Number of participants analyzed = participants with Baseline and Month 6 DTSQ assessment. Missing data imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 346 | 359
units on a scale | 3.05 (0.448) | 3.61 (0.440)

11. Secondary Outcome: Percentage of Participants With Hypoglycemia (All and Nocturnal) Events From Baseline to Month 12
Description: Hypoglycemia events were Severe hypoglycemia (an event that required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions); Documented symptomatic hypoglycemia (typical symptoms of hypoglycemia with plasma glucose level of <=3.9 mmol/L [70 mg/dL]); Asymptomatic hypoglycemia (no typical symptoms of hypoglycemia but plasma glucose level <=3.9 mmol/L); Probable symptomatic hypoglycemia (an event during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination, but was presumably caused by a plasma glucose level <=3.9 mmol/L, symptoms treated with oral carbohydrate without a test of plasma glucose); Relative hypoglycemia (an event during which the person with diabetes reported any of the typical symptoms of hypoglycemia, and interpreted the symptoms as indicative of hypoglycemia, but plasma glucose level >3.9 mmol/L); Severe and/or confirmed a hypoglycemia (plasma glucose <=3.9 mmol/L).
Time Frame: Up to Month 12
Population: Safety population: all participants randomized and exposed to at least one dose of study drug, regardless of the amount of treatment administered. In the event of participants having received treatments different from those assigned according to the randomization schedule, safety analyses were conducted according to treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 403 | 406
percentage of participants
  Any Hypoglycemia Event: All Hypoglycemia | 79.9 | 83.0
  Severe Hypoglycemia: All Hypoglycemia | 1.7 | 1.5
  Documented Symptomatic: All Hypoglycemia | 58.8 | 63.3
  Asymptomatic: All Hypoglycemia | 58.6 | 64.0
  Probable Symptomatic: All Hypoglycemia | 2.7 | 3.4
  Relative: All Hypoglycemia | 7.9 | 12.8
  Severe and/or Confirmed: All Hypoglycemia | 78.4 | 82.0
  Any Hypoglycemia Event: Nocturnal Hypoglycemia | 39.7 | 46.1
  Severe Hypoglycemia: Nocturnal Hypoglycemia | 0.2 | 0.5
  Documented Symptomatic: Nocturnal Hypoglycemia | 29.5 | 34.2
  Asymptomatic: Nocturnal Hypoglycemia | 14.4 | 22.2
  Probable Symptomatic: Nocturnal Hypoglycemia | 1.2 | 1.0
  Relative: Nocturnal Hypoglycemia | 2.2 | 6.4
  Severe and/or Confirmed: Nocturnal Hypoglycemia | 37.5 | 44.6

12. Other Pre Specified Outcome: Change in HbA1c From Month 6 to Month 9
Description: Substudy comparing fixed dosing regimen (every 24 hours) vs. adaptive dosing regimen (every 24 +/- 3 hours) in a subset of participants randomized to HOE901-U300 and treated for 6 months. Only measurements performed before initiation of rescue therapy were considered in the analysis.
Time Frame: Month 6 up to Month 9
Population: mITT substudy population. Number of participants analyzed = participants with Month 6 and Month 9 HbA1c assessment. Analysis was planned to be performed for participants who were receiving HOE901-U300 (Adaptable dosing intervals or Fixed dosing intervals). Missing data imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Groups:
- HOE901-U300: Adaptable Dosing Intervals: HOE901-U300 SC injection once daily for 6 months in combination with oral antidiabetic drug(s). From Month 6 to Month 9 participants received HOE901-U300 once daily at intervals of 24 +/- 3 hours.
- HOE901-U300: Fixed Dosing Intervals: HOE901-U300 SC injection once daily for 12 months in combination with of oral antidiabetic drug(s). From Month 6 up to Month 9 participants received HOE901-U300 once daily every 24 hours.
Arm/Group | HOE901-U300: Adaptable Dosing Intervals | HOE901-U300: Fixed Dosing Intervals
Number analyzed (Participants) | 40 | 37
percentage of hemoglobin | -0.12 (0.151) | -0.25 (0.162)
Statistical Analysis 1: Comparison: HOE901-U300: Adaptable Dosing Intervals vs HOE901-U300: Fixed Dosing Intervals; Analysis was performed using Analysis of covariance (ANCOVA) model with treatment regimen and country as fixed effects and baseline (Month 6) HbA1c value as a covariate; Test type: Superiority or Other; LS Mean Difference = 0.13, 95% CI 2-sided [-0.152 to 0.415], Standard Error of Mean 0.142

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of informed consent form up to study completion regardless of seriousness or relationship to study drug.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from first injection of study drug up to 2 day after the last injection of study drug). Analysis was done on safety population.
Arm/Group | HOE901-U300 | LANTUS
Serious Adverse Events (participants affected / at risk) | 30/403 | 30/406
Other Adverse Events (participants affected / at risk) | 106/403 | 96/406
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HOE901-U300 (N=403) | LANTUS (N=406)
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Nodal rhythm (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Hepatic echinococciasis (Infections and infestations) | 0 | 1
Infected bites (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Superinfection (Infections and infestations) | 1 | 0
Tuberculous pleurisy (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 3
Wound infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Gastroparesis postoperative (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 3
Calculus urinary (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Angiopathy (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HOE901-U300 (N=403) | LANTUS (N=406)
Bronchitis (Infections and infestations) | 25 | 23
Nasopharyngitis (Infections and infestations) | 49 | 31
Upper respiratory tract infection (Infections and infestations) | 23 | 35
Headache (Nervous system disorders) | 27 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.